CLINICAL TRIAL: NCT06225687
Title: The Effect of Heat Application on Gastrointestinal System Functions in Patients Receiving Continuous Enteral Nutrition
Brief Title: Heat Application on Gastrointestinal System Functions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Özlem Ceyhan, Assoc.Prof., TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HeatAppGastro
Record Dates: First submitted 2023-11-28; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Enteral Nutrition; Gastrointestinal System--Abnormalities
Keywords: Enteral Nutrition; Heat Application; Gastrointestinal System Functions; Continuous Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heat Application (Experimental): Heat will be applied to the abdominal/lumbar area for 15 minutes.
  Interventions: Other: Heat Application
- Control Group (No Intervention): No intervention will be made.

INTERVENTIONS:
Other: Heat Application — The researcher will conduct daily measurements of gastric residual volume (GRV) and abdominal circumference, listen to bowel sounds, and assess distension from the first day of enteral nutrition initiation. Additionally, they will record the frequency of vomiting/defecation. Subsequently, a 15-minute hot application will be applied to the abdominal/lumbar region.
  Arms: Heat Application

SUMMARY:
Complications related to the gastrointestinal system can occur in patients receiving enteral nutrition. These complications may include nausea, vomiting, diarrhea, constipation, decreased bowel sounds, abdominal distension, increased gastric residual volume, and abdominal pain. To prevent and treat food intolerance, as well as to increase gastric emptying, the use of prokinetic agents is often preferred. However, these drugs have various side effects, such as abdominal cramps, allergies, bronchospasm, cardiac issues, and pancreatic disorders. One non-pharmacological method that can be applied to increase bowel motility and reduce abdominal distension and constipation is heat application. The aim of this study is to determine the effect of heat application to the abdominal and lumbar regions, using a hot water bag, on gastrointestinal system functions in patients receiving continuous enteral nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Intensive care unit patients
* Individuals aged 18 and above
* Patients receiving enteral nutrition via nasogastric tube
* Patients on the first day of enteral nutrition
* Those receiving standard enteral nutrition solution
* Patients without wounds in the abdominal region
* Individuals who have not undergone abdominal surgery in the last 6 months
* Patients not undergoing radiation/chemotherapy
* Those with a high-output fistula without ileus problems
* Patients without diarrhea and constipation
* Patients with a Glasgow Coma Scale (GKS) > 3
* Those with an APACHE II score > 16
* Patients not taking prokinetic agents
* Patients not taking laxative medications
* Patients without any contraindications for the application of heat, such as neuropathy (to be determined in consultation with the primary doctor).

Exclusion Criteria:

* Patients in whom enteral nutrition is discontinued during the study
* Patients transitioning to a product other than the standard one in enteral nutrition
* Patients who temporarily pause enteral nutrition
* Patients who have started prokinetic agents
* The study will be terminated in patients who have started taking laxative medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Gastric residual volume | 7 days
  GRV measurement will be made 30 minutes after stopping feeding. It will be evaluated before and after application.
Abdominal Distension | 7 days
  Abdominal distension will be assessed 30 minutes after stopping feeding. The palpation method will be used. Additionally, abdominal circumference will be measured with a tape measure. Evaluation will be made before and after the intervention.
Bowel sounds | 7 days
  Bowel sounds should be evaluated 30 minutes after stopping feeding. Bowel sounds are listened to with a stethoscope for one minute. It will be evaluated before and after the intervention.

SECONDARY OUTCOMES:
Defecation Patterns | 7 days
  measure defecation frequency and nature
Vomiting | 7 days
  The number of vomitings during the day is recorded

REFERENCES:
- [Background] Dehghan M, Fatehi Poor A, Mehdipour-Rabori R, Ahmadinejad M. Effect of abdominal massage on prevention of aspiration in intubated and enterally fed patients: A randomized controlled trial. J Complement Integr Med. 2020 Sep 23;17(3). doi: 10.1515/jcim-2017-0124. PMID 31710593
- [Background] Zhang W, Zhou W, Kong Y, Li Q, Huang X, Zhao B, Su H, Chen S, Shen X, Qiu Z. The effect of abdominal massage on enteral nutrition tolerance in patients on mechanical ventilation: A Randomized Controlled Study. Intensive Crit Care Nurs. 2023 Apr;75:103371. doi: 10.1016/j.iccn.2022.103371. Epub 2022 Dec 15. PMID 36528462
- [Background] Uysal N, Eser I, Akpinar H. The effect of abdominal massage on gastric residual volume: a randomized controlled trial. Gastroenterol Nurs. 2012 Mar-Apr;35(2):117-23. doi: 10.1097/SGA.0b013e31824c235a. PMID 22472671
- [Background] Makino Y, Choe MA. Effects of Hot Packs on Small-Intestinal Motility Measured by Doppler Ultrasound and Subjective Feelings in Normal Adults. Gastroenterol Nurs. 2017 Jul/Aug;40(4):279-286. doi: 10.1097/SGA.0000000000000222. PMID 28746113